# ClinicalTrials.gov Study Document

**Official Study Title:** The O2-PRBC. That study on the use of Hemanext One RBC Storage System for blood transfusion support in transfusion-dependent that the study of the use of Hemanext One RBC Storage System for blood transfusion support in transfusion-dependent that the study of the use of Hemanext One RBC Storage System for blood transfusion support in transfusion-dependent that the study of the use of Hemanext One RBC Storage System for blood transfusion support in transfusion-dependent that the study of the use of Hemanext One RBC Storage System for blood transfusion support in transfusion-dependent that the use of Hemanext One RBC Storage System for blood transfusion support in transfusi

NCT Number: Pending

Document Type: Study Protocol and Statistical Analysis Plan Document

**Date:** NOV 2025

# Study/Protocol Title: The αO2-PRBC.Thal study on the use of Hemanext One® RBC Storage System for blood transfusion support on transfusion-dependent thalassemia

#### Introduction

Patients with transfusion dependence thalassemia (TDT) are regularly transfused every two to four weeks. Their long-term survival and quality of health is dependent on the quality of the transfused blood. TDT patients experience significant problems and organ dysfunction due to chronic anemia, chronic iron overload as well as long life use of different medications, like iron chelators. TDT patients usually receive 2-4 units of red blood cells (RBC) (each unit: 250300ml), per month.

RBCs storage processing aims to preserve the RBCs' properties. Long-term storage leads to donor-dependent biochemical and morphological changes in RBCs collectively termed as "storage lesions". Transfusion of stored RBCs for more than 1 to 2 weeks is associated with increased post-transfusion mortality rates [1-4]. Therefore, there is a need for developing optimized processing and storage conditions. Considering the primary functional role of RBCs, which is oxygen transport and exchange, focusing on these processes might be a potential way for improving storage quality [1,5].

RBCs' "storage lesions" have recently been correlated with metabolic reprogramming [6]. Dysregulation of RBCs' homeostasis disrupts structural lipids and proteins, resulting in progressive pathological alterations in RBC morphology, and downregulates RBCs' survival post-transfusion [6]. "Storage lesions" represent a wide spectrum of RBCs' deformities being associated with oxidative damage, manifesting as post-translational changes in proteins (e.g., hemoglobin, peroxiredoxin 2, anion exchanger 1, catalase, pyruvate kinase, glucose 6phosphate dehydrogenase) and depletion of redox metabolites (e.g., glutathione) [7-13]. Glycolytic enzymes, especially glyceraldehyde 3-phosphate dehydrogenase (GADPH), have been shown in vitro to mediate this process; oxygen is considered to modulate the competitive binding of glycolytic enzymes and deoxyhemoglobin with N-terminal cytosolic domains [14]. Specifically, GADPH, is linked to the depletion of 2,3-diphosphoglycerate (2,3-DPG) during the first 2 weeks of storage [3,9,15-17]. Oxygen saturation levels are considered to modulate the competitive binding of GADPH and deoxyhemoglobin with N-terminal cytosolic domains [14]. Under pro-oxidant conditions, hemoglobin turns into its oxygenated substance decreasing its binding affinity, while GADPH, migrates to binding sited of the nearby structural proteins. Ectopic localization of GADPH to the membrane and binding with structural proteins, has been associated with loss of activity, blocking glycolysis, and causing various morphologic and functionality defects on the binding proteins [14].

Studies have shown that RBCs stored under hypoxic conditions preserved faster O<sub>2</sub> kinetics compared with the standard storage protocols, with this difference being reported in the first 35 days of storage; that is, the longest permissible shelf-life of blood in the United Kingdom and many European countries [1]. In clinical practice, the median storage duration of transfused units is 21 days. The effects on O<sub>2</sub> after RBCs' storage in hypoxic conditions are similar to the ones of biochemical rejuvenation following standard storage – however RBCs' storage in hypoxic conditions presents advantages in terms of easier clinical use, as it can be conducted on units in bulk and before dispatch to hospitals [1].

The Hemanext ONE RBC Processing and Storage system limits oxygen, the fuel for oxidative damage, thus, providing a higher quality RBCs. It has the potential to benefit all patients requiring transfusion for chronic conditions such as thalassemia, sickle cell disease (SCD), and myelodysplastic syndromes (MDS), as well as those in need of critical transfusions during post-traumatic surgery and other medical procedures [18-26]. Hemanext ONE creates hypoxic RBCs, RBCs that have been processed to reduce oxygen and carbon dioxide content of RBCs and to maintain this level throughout storage up to 42 days. Hypoxic RBCs have demonstrated positive impacts on multiple in vitro metrics of RBC quality in preclinical studies. Clinical studies are underway to determine the impact of hypoxic RBCs on patient outcomes and estimate potential cost savings from expected improvements in care and reductions in transfusion volumes.

Hemanext ONE has been granted marketing authorization for commercial distribution via the De Novo process by the U.S. Food & Drug Administration. In Europe, Hemanext ONE is CE marked which allows the medical device to be placed in the market in the European Economic Area (EEA).

Hemanext ONE has not been studied in chronically transfused patients like thalassemia. It is imperative to establish the safety and the efficacy, especially in regard to required quantity of blood transfusion prepared with the Hemanext ONE processing, before its general application to sensitive groups of patients like TDT. In this respect, there are many issues to be investigated, like long-term biochemical results and changes in the primary physiological function of RBCs in thalassemic recipients.

The aim of our study is to investigate whether RBCs' storage under hypoxic conditions is at least non inferior to standard conditions in providing transfusion support to TDT patients without increasing the transfusion burden, the degree of hemolysis and of metabolic disturbances, and the rate of iron and erythropoiesis, while improving our patients' quality of life (QOL).

#### **Objectives**

- To validate the feasibility of applying the Hemanext ONE processing and storage of blood units in the routine care of transfusion dependent thalassemic (TDT) patients
- To evaluate the safety of Hemanext ONE in TDT
- To evaluate the changes in transfusion burden when using the Hemanext ONE system
- To evaluate changes in surrogate markers of metabolism, hemolysis, iron overload and erythropoiesis, when using the Hemanext ONE system
- To assess QOL changes

### **Hypothesis**

The hypothesis is that using the hemanext one process is able to provide transfusion support to TDT patients without increasing the transfusion burden, the degree of hemolysis and metabolic disturbances, and the rate of iron and erythropoiesis.

# **Primary Endpoint**

Changes from baseline in RBC transfusion burden. Significant changes are defined as a difference of >20% from baseline, corresponding to at least 1 unit/24weeks.

# **Secondary Endpoints**

- Changes from baseline in pre-transfusion hemoglobin
- Changes on mean total Hb mass
- Changes from baseline in metabolic markers
- Changes from baseline in other markers of hemolysis and erythropoiesis
- Changes in OOL
- Overall changes from baseline in markers of iron overload
- Type, frequency, severity, seriousness of AEs and relationship of AEs to Hemanext. AEs of interest include hemolytic reactions and

#### METHODOLOGY

#### **Patients**

TDT patients followed at the Thalassemia Unit either of the First Dept of Pediatrics NKUA or at the LAIKON General Hospital and fulfilling the following criteria will be invited to participate in the study.

#### **Inclusion Criteria**

Subjects must satisfy the following criteria to be enrolled in the study:

- 1. Subject is  $\geq$  18 years of age at the time of signing the informed consent form (ICF).
- 2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
- 3. Subject has documented diagnosis of  $\beta$  transfusion dependent thalassemia, defined as ect:  $\geq 6$  RBC units/24 weeks and no transfusion-free period for  $\geq 42$  days during the 24 weeks prior enrollment.
- 4. Transfusion history (including units or cc) for at least 6 months prior to enrollment needs to be available.
- 5. Subject is on chelation therapy and a fairly stable dose for at least 6 months prior to enrollment.
- 6. Chronic therapies (including hydroxyurea) are allowed as long as the medication dose has been stable for at least 6 months prior to enrollment.
- 7. Having been exposed to PRBC transfusions prepared with the Hemanext One processing system

#### **Exclusion Criteria**

The presence of any of the following will exclude a subject from enrollment:

- 1. Subject has currently or has a history of any significant medical condition, laboratory abnormality, or psychiatric illness.
- 2. Subject has had positive Coombs (antiglobulin) test anytime during the 6 months prior to enrollment.
- 3. Subject is scheduled to undergo or has recently (in the last 6 months) undergone splenectomy.
- 4. Use of luspatercept during the period of 6 months prior to enrollment and during the trial is not allowed.

5. Participation in an interventional clinical trial or use of experimental medications during the period of 6 months prior to enrollment and during the trial is not allowed.

#### Methods

The trial will consist of two phases.

# • Baseline phase (retrospective or prospective)

The baseline phase consists of 12 weeks, evaluated retrospectively or prospectively, just prior or after receiving Hemanext transfusion. During this phase, the patients are expected to have received packed red blood cells (PRBC) processed using standard method. The phase will be used to establish their baseline transfusion and hematologic characteristics. Baseline values will be derived from this phase.

#### • Treatment Phase

The treatment phase will last for at least 3 months, during which patients will continue receiving PRBCs prepared using the Hemanext methodology. This phase will continue for as long as the patient receives Hemanext-prepared PRBC transfusions and may be extended until the data cut-off date. The data cut-off date is defined as the time point when data have been collected for at least 3 months from all patients included in the study. Each patient must sign the Informed Consent Form before any data collection begins.

HEMANEXT ONE process and store CP2D/AS-3 Red Blood Cells, Leukocytes Reduced (LR RBC) that have been prepared within the standard 8-hour hold time. Processing must be initiated within 8 hours of collection and completed within 12 hours of collection. The Red Blood Cells must be processed at room temperature (20-26°C). The HEMANEXT ONE system limits O<sub>2</sub> and CO<sub>2</sub> levels in the storage environment. Red Blood Cells Leukocytes Reduced, O<sub>2</sub>/ CO<sub>2</sub> Reduced may be stored for up to 42 days at 1-6°C. HEMANEXT ONE is used for volumes no greater than 350 mL of LR RBC.

#### **Transfusion Burden**

As this is the primary end point, the transfusion burden should be calculated based on cc/kg. Number of blood units could also be registered and if available hematocrit of the PRBC's. Baseline values will be based on the baseline phase.

# **Transfusion Efficacy**

To evaluate further the efficacy of the transfusion, the mean total Hb mass will be calculated based on Nadler's formula for blood volume, as follows:

For males = 
$$(0.3669 \times height(m)^3 + 0.03219 \times body weight(kg) + 0.6041) \times mean Hb (g/L)$$

For females = 
$$(0.3561 \times height(m)^3 + 0.03308 \times body weight(kg) + 0.1833) \times mean Hb (g/L)$$

Mean Hemoglobin calculated as the sum of the values of the mean hemoglobin between two measurements multiply by the  $\times \frac{(days\ between\ 2\ measurement)}{(total\ observation\ period)}$ 

# Analyses

Different analysis will be evaluated as per standard follow up protocols for these patients. Samples for further exploratory analyses will be collected and stored

Samples collection and timepoints

| Visit Week: | | riod | | | Treatment Phase | | | | | | | | | Open-Label<br>Extension<br>Period | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 1 | | | | | | 13 | 14 | | | | | | | | 38 | Till LPLV |
| Study Day: | 1 | | | | | | 85 | 92 | | | | | | | | 260 | |
| Transfusion Day: | | | | | | | | | | | | | | | | | |
| Informed consent | | | | | | | | X | | | | | | | | | |
| Demographics <sup>2</sup> | X | | | | | | | | | | | | | | | | |
| Eligibility | X | | | | | | | | | | | | | | | | |
| Medical and surgical history | X | | | | | | | X | | | | | | | | X | |
| Transfused PRBC cc/kg – units | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Medications | X | | | | | | | X | | | | | | | | X | X |
| Vital signs | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Hematology, including reticulocytes | X | | | | | | | X | | • | | X | | | | | |
| Serum chemistry | X | As per standard evaluation | | | | | | X | | | | | | | | | As per standard practice |
| Liver function tests | X | | | | | | | X | | As per standard | | | | | | X | As per standard practice |
| Lipid panel | X | | | | | | | X | | evaluation | | | | | | | As per<br>standard<br>practice |
| Iron panel | X | | | | | | | X | | | | | | | | X | Q 3months |
| QOL | | | | | | | | X | | | | | | | | X | At last visit |

| Blood sample for<br>exploratory<br>disease<br>parameters | | X | | | | | X | At last visit |
|---|---|---|---|---|---|---|---|---|
| Adverse events<br>and serious<br>adverse events | X | | X | (con | tinuc | ous) | | |

LV: last visit with Hemanext

LPLV: Last patient last visit during treatment phase

Hematology includes complete blood count with differential, HCT, Hb, RBC count, absolute reticulocyte count, percent reticulocyte count, MCV, MCH, MCHC, RDW, WBC count with differential, and platelet count.

Serum chemistry includes sodium, potassium, chloride, calcium, magnesium, phosphorus, carbon dioxide or bicarbonate, albumin, total protein, glucose, BUN or urea, creatinine, and uric acid.

Liver function tests include LDH, ALP, ALT, AST, and bilirubin (total, direct, and indirect). Lipid panel includes total cholesterol, LDL-C, HDL-C, and triglycerides; samples will be collected after an overnight fast. Iron panel may include iron, serum ferritin, total iron binding capacity, or transferrin saturation.

#### **Statistical Method:**

For continuous parameters, summary statistics will include the number of subjects, mean, standard deviation, quartiles, minimum and maximum, and the 95% confidence interval of the mean (if appropriate). For categorical parameters, summary statistics will include counts, percentages, and the 95% confidence interval of the percentages (if appropriate) in each category.

Based on analysis on random patients from our unit, the standard deviation (SD) of transfusion burden (annual consumption in cc/kg/year) was estimated at 22.8. The non-inferiority limit was set at 15%. For a power of 90%, 25 participants are required. Assuming a drop-out rate of 10%, the target enrollment will be at least 28 patients.

An interim analysis will be performed when half of the expected enrolled patients (the 15<sup>th</sup> patient) have reached week 12 of the treatment phase.

#### References

- 1. Rabcuka J, Blonski S, Meli A, et al. Metabolic reprogramming under hypoxic storage preserves faster oxygen unloading from stored red blood cells. *Blood Adv.* 2022;6(18):5415-5428. doi: 10.1182/bloodadvances.2022007774
- 2. Bennett-Guerrero E, Veldman TH, Doctor A, et al.. Evolution of adverse changes in stored RBCs. *Proc Natl Acad Sci USA*.2007;104(43): 17063-17068.
- 3. Hess JR. Measures of stored red blood cell quality. Vox Sang. 2014;107(1):1-9.
- 4. Roussel C, Dussiot M, Marin M, et al.. Spherocytic shift of red blood cells during storage provides a quantitative whole cell-based marker of the storage lesion. *Transfusion*. 2017;57(4):1007-1018.
- 5. Peter Klinken S. Red blood cells. Int J Biochem Cell Biol. 2002 Dec;34(12):1513-8. doi: 10.1016/s1357-2725(02)00087-0. PMID: 12379271.
- 6. Reisz JA, Wither MJ et al. Oxidative modifications of glyceraldehyde 3-phosphate dehydrogenase regulate metabolic reprogramming of stored red blood cells. 2016;128(12): e32-42.
- 7. Rinalducci, Sara, Cristina Marrocco, and Lello Zolla. "Thiol-based regulation of glyceraldehyde-3-phosphate dehydrogenase in blood bank—stored red blood cells: a strategy to counteract oxidative stress." *Transfusion* 55, no. 3 (2015): 499-506.
- 8. Dandekar, Thomas, Astrid Fieselmann, Saman Majeed, and Zeeshan Ahmed. "Software applications toward quantitative metabolic flux analysis and modeling." *Briefings in bioinformatics* 15, no. 1 (2014): 91-107.
- 9. D'Alessandro, Angelo, Monika Dzieciatkowska, Ryan C. Hill, and Kirk C. Hansen. "Supernatant protein biomarkers of red blood cell storage hemolysis as determined through an absolute quantification proteomics technology." *Transfusion*56, no. 6 (2016): 1329-1339.
- 10. Chouchani, Edward T., Andrew M. James, Ian M. Fearnley, Kathryn S. Lilley, and Michael P. Murphy. "Proteomic approaches to the characterization of protein thiol modification." *Current opinion in chemical biology* 15, no. 1 (2011): 120-128.
- 11. Clasquin, Michelle F., Eugene Melamud, and Joshua D. Rabinowitz. "LC-MS data processing with MAVEN: a metabolomic analysis and visualization engine." *Current protocols in bioinformatics* 37, no. 1 (2012): 14-11.
- 12. Nemkov, Travis, Angelo D'Alessandro, and Kirk C. Hansen. "Three-minute method for amino acid analysis by UHPLC and high-resolution quadrupole orbitrap mass spectrometry." *Amino acids* 47 (2015): 2345-2357.
- 13. Dzieciatkowska, Monika, Ryan Hill, and Kirk C. Hansen. "GeLC-MS/MS analysis of complex protein mixtures." *Shotgun Proteomics: Methods and Protocols* (2014): 5366.
- 14. Julie A. Reisz, Matthew J. Wither, Monika Dzieciatkowska, Travis Nemkov, Aaron Issaian, Tatsuro Yoshida, Andrew J. Dunham, Ryan C. Hill, Kirk C. Hansen, Angelo D'Alessandro, Oxidative modifications of glyceraldehyde 3-phosphate dehydrogenase regulate metabolic reprogramming of stored red blood cells, Blood, Volume 128, Issue 12, 2016, ISSN 0006-4971, https://doi.org/10.1182/blood-2016-05-714816.
- 15. van der Meer PF, Cancelas JA, Cardigan R, et al.; BEST Collaborative . Evaluation of overnight hold of whole blood at room temperature before component processing: effect of red blood cell (RBC) additive solutions on in vitro RBC measures. *Transfusion*. 2011;51(suppl 1):15S-24S.

- 16. Wilsher C, Garwood M, Sutherland J, Turner C, Cardigan R. The effect of storing whole blood at 22 degrees C for up to 24 hours with and without rapid cooling on the quality of red cell concentrates and fresh-frozen plasma. *Transfusion*.2008;48(11):2338-2347.
- 17. Dern RJ, Brewer GJ, Wiorkowski JJ. Studies on the preservation of human blood. II. The relationship of erythrocyte adenosine triphosphate levels and other in vitro measures to red cell storageability. *J Lab Clin Med.* 1967;69(6):968-978.
- 18. HEMANEXT ONE® (Blood container set used to process and store CP2D/AS-3 Red Blood Cells, Leukocytes Reduced, and O<sub>2</sub>/CO<sub>2</sub> Reduced) [US Instructions for Use]. Lexington, MA: Hemanext Inc.
- 19. Farmakis D, Porter J, Taher A, et al. 2021 Thalassemia International Federation Guidelines for the management of transfusion-dependent thalassemia. 2022;6:8.
- 20. Chou S, Alsawas M, Fasano R, et al. American Society of Hematology 2020 guidelines for sickle cell disease: transfusion support. *Blood Adv.* 2020;4:2.
- 21. Germing U, Oliva E, Hiwase D, and Almeida A. Treatment of anemia in transfusiondependent and non-transfusion-dependent lower-risk MDS: current and emerging strategies. 2019;3(6). doi: 10.1097/HS9.000000000000314
- 22. American College of Surgeons. ACS TQIP massive transfusion in trauma guidelines. *ACS TQIP*. 2014; https://www.facs.org/media/zcjdtrd1/transfusion guildelines.pdf.
- 23. Yoshida T, Blair A, D'Alessandro A, et al. Enhancing uniformity and overall quality of red cell concentrate with anaerobic storage. *Blood Transfus*. 2017;15(2):172-81.
- 24. Yoshida T, McMahon E, Croxon H, et al. The oxygen saturation of red blood cell concentrates: The basis for a novel index of red cell oxidative stress. Transfusion. 2022;62(1):183-193. doi: 10.1111/trf.16715.
- 25. Reikvam H, Hetland G, Ezligini F, et al. Safety of hypoxic red blood cell administration in patients with transfusion-dependent hematological malignancies: An interim analysis. *Transfus Apher Sci.* 2023; doi: 10.1016/j.transci.2023.103755.